CLINICAL TRIAL: NCT01520389
Title: A Phase 1 and Pharmacologic Study of MM-151 in Patients With Refractory Advanced Solid Tumors
Brief Title: Safety Study of the Drug MM-151 in Patients With Advanced Solid Tumors Resisting Ordinary Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merrimack Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM-151-01-01-01
Record Dates: First submitted 2012-01-13; First posted 2012-01-30 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Advanced Solid Tumors; Colorectal Cancer; Squamous Cell Head and Neck Cancer; Non Small Cell Lung Cancer; Triple Negative Breast Cancer
Keywords: cancer; solid tumors; oncology; Phase I; EGFR; EGF receptor (ErbB1); irinotecan
MeSH Terms: conditions — Colorectal Neoplasms; Head and Neck Neoplasms; Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms; Neoplasms | interventions — MM-151; Irinotecan

ARMS (3):
- MM-151 Dose Escalation (Experimental): MM-151 Dose escalation frequency - once weekly, once every two weeks, once every three weeks
  Interventions: Drug: MM-151
- MM-151 Expansion in KRAS wild type colorectal cancer (Experimental): MM-151 given weekly
  Interventions: Drug: MM-151
- MM-151 + irinotecan (Experimental): MM-151 given weekly, irinotecan 180 mg/m2 given once every two weeks
  Interventions: Drug: MM-151 + irinotecan

INTERVENTIONS:
Drug: MM-151 — MM-151
  Arms: MM-151 Dose Escalation; MM-151 Expansion in KRAS wild type colorectal cancer
Drug: MM-151 + irinotecan — MM-151 + irinotecan
  Other Names: camptosar
  Arms: MM-151 + irinotecan

SUMMARY:
This study is a Phase 1 and pharmacologic open-labeled dose-escalation trial using a "3+3" design, evaluating MM-151 at varying dose levels and frequencies, and subsequently in combination with irinotecan.

DETAILED DESCRIPTION:
This study is a Phase 1 and pharmacologic open-labeled dose-escalation trial using a "3+3" design exploring weekly, bi-weekly, and tri-weekly dosing schedules. Successive MM-151 monotherapy cohorts of three or more patients will be treated at escalating doses until a maximum tolerated dose is identified, and subsequently in combination with irinotecan. The study consists of three parts as follows: MM-151 monotherapy dose escalation (Part 1); MM-151 monotherapy expansion cohort in cetuximab-refractory colorectal cancer (Part 2); MM-151 + irinotecan dose escalation (Part 3). It is expected that approximately 4 study sites will participate.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed advanced malignant solid tumor that has recurred or progressed following standard therapy, or that has not responded to standard therapy, or for which there is no standard therapy, or who are not candidates for standard therapy
* Patients must be > 18 years of age
* Patients of their legal representatives must be able to understand and sign an informed consent form
* Patients must have evaluable or measurable tumor(s)
* Patients must be recovered from the effects of any prior surgery, radiotherapy or other antineoplastic therapy. Up to CTCAE Grade 1 is acceptable for patients with known peripheral neuropathy
* Women of childbearing potential as well as fertile men and their partners must agree to abstain from sexual intercourse or to use an effective form of contraception during the study and for 90 days following the last dose of MM-151 (an effective form of contraception is an oral contraceptive or a double barrier method)

Exclusion Criteria:

* Patients for whom potentially curative antineoplastic therapy is available
* Patients who are pregnant or lactating
* Patients with an active infection or with an unexplained fever > 38.5°C during screening visits or on the first scheduled day of dosing. (At the discretion of the investigator, patients with tumor fever may be enrolled.)
* Patients with untreated and/or symptomatic CNS malignancies (primary or metastatic); patients with CNS metastases who have undergone surgery or radiotherapy, whose disease is stable, and who have been on a stable dose of corticosteroids for at least 2 weeks prior to the first scheduled day of dosing will be eligible for the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Phase II dose of MM-151 alone and in combination with irinotecan based either on the maximum tolerated dose (MTD) or maximum dose of 18 mg/kg in patients with advanced solid malignancies. | Two years

SECONDARY OUTCOMES:
Number of dose limiting toxicities (DLTs) within a cohort | 2 years
Adverse event profile of MM-151 alone and in combination with irinotecan | 2 years
Objective response to MM-151 alone and in combination with irinotecan based on RECIST | 2 years

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Colorado Denver, Aurora, Colorado
  - Horizon Oncology Research, Inc., Lafayette, Indiana
  - Roswell Park Cancer Institute, Buffalo, New York
  - South Texas Accelerated Research Therapeutics, LLC (START), San Antonio, Texas